CLINICAL TRIAL: NCT07130422
Title: Incidence and Risk Factors of Surgical Site Infections After Coronary Artery Bypass Grafting Surgery: A Prospective Observational Study in a Tertiary Care Center in Nepal
Brief Title: Incidence and Risk Factors of Surgical Site Infections After Coronary Artery Bypass Grafting Surgery
Status: Completed | Type: Observational
Sponsor: Maharajgunj Medical Campus (Other)
Responsible Party: Principal Investigator, Prajjwol Luitel, Principal Investigator, Maharajgunj Medical Campus
Other Study IDs: 588(6-11)E2.079/080
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: CABG

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CABG surgery
  Interventions: Procedure: CABG surgery

INTERVENTIONS:
Procedure: CABG surgery — CABG surgery

SUMMARY:
The burden of coronary artery disease (CAD) is increasing in the Nepalese population. Coronary artery bypass grafting (CABG) remains one of the most frequently performed surgical interventions for the management of advanced CAD. Despite this, there is a paucity of data regarding the incidence and determinants of surgical site infections (SSIs) following CABG in the Nepalese context. This study aimed to determine the incidence of SSIs after CABG surgery in the Nepalese population.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Undergoing isolated coronary artery bypass graft (CABG) surgery
* Elective surgical cases

Exclusion Criteria:

* CABG performed in combination with other cardiac procedures (e.g., valve surgery, aortic aneurysm repair, congenital heart surgery)
* Known allergy to penicillin or cephalosporins
* Refusal to provide informed consent
* Loss to follow-up within 30 days after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted at Manmohan Cardio Thoracic Vascular and Transplant Center (MCVTC), a national tertiary referral center in Nepal performing over 20% of the country's cardiac surgeries. Using convenience sampling, adults (≥18 years) undergoing elective, isolated CABG were included. Patients having combined cardiac procedures, penicillin/cephalosporin allergy, refusal of consent, or loss to follow-up within 30 days were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Surgical Site Infection (SSI) Following Coronary Artery Bypass Grafting (CABG) | 30 days post-CABG
  The study aims to assess the proportion of patients developing surgical site infections within the first 30 days after undergoing coronary artery bypass graft surgery. SSIs will be identified based on standardized diagnostic criteria, and cases will be classified according to infection depth and site. Data collection will include clinical examination findings, laboratory results, and relevant imaging, ensuring comprehensive identification and categorization of infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Nepal, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Undecided